## **Informed Consent and Child Assent**

Official Title of the Study: Knowledge Accessibility and Availability in Forming Knowledge-to-Text

Inferences among Middle Grade Readers

NCT number: NCT03782012

Date of the Document: 27 August 2023

## The Knowledge Project

Dear Parent or Guardian:

Dr. Amy Barth at Buena Vista University studies how to improve the reading outcomes of students in middle school. This study will look at how students combine information from print with their knowledge of the topic. This study will help identify how classroom instruction can be improved.

Because of the importance of this research, Storm Lake Middle School is partnering with Dr. Barth. Beginning in the fall, your student will complete some tests that measure different reading skills and factors that impact reading. Your student will also learn some facts about a planet, and then be tested on how well they remember the facts, use the facts during reading, and remember the facts one week later. All tests will be administered by a highly trained student from Buena Vista University.

No risks are associated with this research study.

Your student and future students may benefit from this study because scientists and teachers will learn how to build knowledge before reading and help students think deeply about different texts.

Dr. Barth will keep a record of your student's performance in a secure database. Your student will not be identified by their name. Only Dr. Barth and Mr. Slight will know the identity of all participants. All data is confidential.

You may withdraw your student at any time without penalty.

If you have any questions or concerns, please talk to Mr. Slight or Dr. Barth.

If you do not want your student to participate, check the box below, write your student's name and your name on the lines below, and return this form to the Storm Lake Middle School Office.

Respectfully,

Amy E. Barth, Ph.D., CCC-SLP

Assistant Professor, Literacy

Mr. J.B. Slight

Principal, Storm Lake Middle School

I do not want to participate.

\_\_\_\_\_Student Name
Parent Signature

| Introduction to Student ar | d Child Assent: |
|---|---|
| help middle school studenthat we can help others im will seem very easy, while passage. The information any time during the testing | I work for the Buena Vista University. We are conducting a research study to as become better readers. We are asking students like you to work on this project so prove their reading skills. I will be asking you some questions and problems that others will seem hard. You will read passages and answers questions about the you give me will in no way affect your grade, it is for research purposes only. If at you are uncomfortable and would like to talk with your school counselor, you may estions? Do you agree to participate in this research study? |
| Student's Signature: | |